CLINICAL TRIAL: NCT07212621
Title: Effects of Three Different Pilates Methods on Pelvic Floor Muscle Function
Brief Title: Relationship Between Trunk Muscles and Pelvic Floor Strength
Acronym: PelvicFloor
Status: Completed | Type: Observational
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Burçin Uğur Tosun, Principal Investigator PhD Physiotherapist Burcin Ugur Tosun, Eastern Mediterranean University
Other Study IDs: PelvicFloorAssessmentAndRehab
Record Dates: First submitted 2025-09-23; First posted 2025-10-08 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Pelvic Floor Muscle Weakness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In recent years, the pelvic floor has emerged as a focal point for both academic research and clinical practice. This dynamic, hammock-like structure, comprising the pubococcygeus, iliococcygeus, coccygeus, and puborectalis muscles, provides essential support to the uterus, bladder, and rectum. This study aims to investigate the relationship between core endurance and pelvic floor muscle strength, shedding light on their interdependent roles in therapeutic outcomes.This study aimed to investigate the relationship between core endurance and pelvic floor muscle strength and endurance in healthy women, commencing on May to June 2025.

DETAILED DESCRIPTION:
In recent years, the pelvic floor has emerged as a focal point for both academic research and clinical practice. This dynamic, hammock-like structure, comprising the pubococcygeus, iliococcygeus, coccygeus, and puborectalis muscles, provides essential support to the uterus, bladder, and rectum. The pelvic floor plays a critical role in maintaining core stability, ensuring continence, and supporting reproductive health, underscoring its profound functional significance.

The pelvic floor muscles are susceptible to weakening due to various factors, including aging, menopause, obesity, pregnancy, and traumatic childbirth. This compromised muscle integrity is closely associated with clinical conditions such as urinary incontinence and pelvic organ prolapse, underscoring the significant implications of impaired pelvic floor function.

The pelvic floor muscles, multifidus, transversus abdominis, and diaphragm collectively form a protective 'capsule' surrounding the abdominal and pelvic organs. The pelvic floor acts as the inferior boundary, with the abdominal muscles forming the lateral walls. Their coordinated contraction enhances spinal and pelvic stability, highlighting their critical, integrated role in core support.

Kegel originally posited that the pelvic floor and abdominal muscles contract concurrently. Subsequent electromyography (EMG) studies have substantiated this, demonstrating a clear relationship between the pelvic floor muscles and both the transversus abdominis and internal oblique muscles. Additionally, Bo et al. documented co-activation of the pelvic floor and abdominal muscles during arm elevation and overhead tasks, further illuminating their functional interdependence. Richardson et al. identified a strong correlation between pelvic floor and abdominal muscle activity, observed through palpation-detected spasms in the abdominal muscles of women. In a systematic review, Bo et al. further noted that this synergy between the pelvic floor and abdominal muscles may weaken or vanish entirely when pelvic floor muscle strength declines, highlighting the interdependence of these structures.

This study aims to investigate the relationship between core endurance and pelvic floor muscle strength, shedding light on their interdependent roles in therapeutic outcomes.

Material Method This study aimed to investigate the relationship between core endurance and pelvic floor muscle strength and endurance in healthy women, commencing on May to June 2025. Approval and permission for the study were obtained from the Health Ethics Subcommittee of the Eastern Mediterranean University Scientific Research and Publication Ethics Board.

Assessments were conducted at the Adana Active Life Center Physiotherapy Clinic and the Eastern Mediterranean University Physiotherapy Department in Cyprus. Prior to the study, all participants were informed about its purpose, the assessments to be conducted, and the subject matter, and they voluntarily signed an informed consent form.

Participants This study enrolled 25 healthy women aged 35-50 who had given birth no more than three times and were premenopausal. Inclusion criteria included no chronic diseases, no alcohol or tobacco use, and a sedentary lifestyle. Exclusion criteria were pregnancy and a history of preterm birth.

Assessments At the start of the assessment session, participants' age, weight, and body mass index (BMI), number of births, education level, employment status were measured and recorded on a sociodemographic form. Then strength and endurance measurements were conducted by a trained physiotherapist.

Pelvic Floor Muscle Strength and Endurance: A perineometer (specifications to be confirmed) was used to assess participants in a supine hook-lying position. For strength, participants performed three maximal contractions, with the average pressure recorded. For endurance, 60% of the maximum contraction value was calculated, and participants were instructed to sustain this target pressure, as displayed on the perineometer. The test ended at the onset of fatigue or when contraction strength dropped to 50% of the target, with duration recorded in seconds.

McGill Core Endurance Tests:

Lateral Bridge Test: Participants assumed a side bridge position, supporting themselves on their elbow and feet. After practice attempts, the duration of maintaining this position was recorded in seconds using a stopwatch.

Trunk Flexor Endurance Test: Using the McGill Core Endurance Test Battery, the time participants sustained a flexion position was measured in seconds with a stopwatch.

Trunk Extensor Endurance Test: Participants lay prone, with pelvis, hips, and knees supported on a table, and the upper body extended beyond the table's edge from the pelvis upward. The therapist stabilized the lower extremities, and the time the trunk maintained a horizontal position was recorded in seconds using a stopwatch.

ELIGIBILITY:
Inclusion Criteria:

-Sedentary lifestyle

Exclusion Criteria:

* Women who were pregnant or
* Had a history of preterm birth
* Smokers
* Drinkers
* Chronic diseases

Ages: 18 Years to 50 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Women
Study Population: The study included 60 healthy premenopausal women between the ages of 18 and 50, all of whom had experienced no more than three full-term births.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-08-27 (Actual); Study Completion 2025-08-27 (Actual)

PRIMARY OUTCOMES:
Pelvic Floor Muscle Strength and Endurance: | "At enrollment (one-time measurement)"
  Pelvic floor muscle (PFM) strength and endurance were evaluated using a perineometer (device specifications to be confirmed), with participants positioned in the supine hook-lying posture. For strength assessment, each participant was instructed to perform three maximal voluntary contractions of the pelvic floor muscles. The mean pressure value across the three trials was recorded as the strength score. For endurance assessment, 60% of the participant's maximum contraction value was calculated, and participants were asked to maintain this target pressure, as visualized on the perineometer display. The test was terminated upon the onset of fatigue or when the contraction pressure dropped to 50% of the target value. Endurance was recorded in seconds.

SECONDARY OUTCOMES:
McGill Core Endurance Tests (Trunk Lateral Bridge Test) | At baseline (single assessment at study entry)
  Participants assumed a side bridge position, supporting themselves on their elbow and feet. After practice attempts, the duration of maintaining this position was recorded in seconds using a stopwatch.
  Trunk Flexor Endurance Test: Using the McGill Core Endurance Test Battery, the time participants sustained a flexion position was measured in seconds with a stopwatch.
  Trunk Extensor Endurance Test: Participants lay prone, with pelvis, hips, and knees supported on a table, and the upper body extended beyond the table's edge from the pelvis upward. The therapist stabilized the lower extremities, and the time the trunk maintained a horizontal position was recorded in seconds using a stopwatch.

OTHER OUTCOMES:
McGill Core Endurance Tests (Trunk Flexor Endurance Test) | At baseline (single assessment at study entry)
  Using the McGill Core Endurance Test Battery, participants sustained a trunk flexion position with the back supported at 60° from horizontal. The duration of maintaining this position was measured in seconds with a stopwatch.
McGill Core Endurance Tests (Trunk Extensor Endurance Test) | At baseline (single assessment at study entry)
  Participants lay prone with the pelvis, hips, and knees supported on a table, while the upper body extended beyond the table's edge from the pelvis upward. The lower extremities were stabilized by the therapist. The time the participant maintained the trunk in a horizontal position was measured in seconds using a stopwatch.

CONTACTS AND LOCATIONS:
Overall Officials: Çisel Demiralp, Phd, Principal Investigator — Eastern Mediterrenean Univeristy
Locations (1):
- Eastern Mediterranean University, Famagusta, Cyprus